CLINICAL TRIAL: NCT02084394
Title: Non Invasive Monitoring of Cerebral Blood Flow During and After Cardiopulmonary Bypass to Assess and Compare for the Presence of Delirium in Post Operative Patients (DELIRIUM)
Brief Title: Cerebral Blood Flow During CPB During Cardiac Surgery and the Presence of Post op Delirium
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Ornim Medical (Industry)
Responsible Party: Principal Investigator, Dr Kaushik Mandal, Assistant Professor Division of Cardiac Surgery, Johns Hopkins University
Other Study IDs: NA_0007115
Record Dates: First submitted 2014-02-25; First posted 2014-03-12 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Delirium
Keywords: CBF autoregulation, rSO2,doppler, TCD, delirium,
MeSH Terms: conditions — Delirium; Choroideremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no intervention: Contact with enrolled subjects requires application of ceberal oximetry electrodes and the concommittent ultrasound of the temporal artery. Deemed interventional by JHUIRB but no actual intervention done to subject.

SUMMARY:
Cardiac surgery is associated with multiple events and issues that increase risk for adverse postoperative neurological outcomes including postoperative cognitive dysfunction. The risk for postoperative delirium is generally thought to result from some previous health factors added to the susceptibility of the cardiac surgery process.

DETAILED DESCRIPTION:
Cardiac surgery is associated with multiple perturbations that increase risk for adverse postoperative neurological outcomes including postoperative cognitive dysfunction. These same perturbations likely also increase the risk for postoperative delirium although there are little data that have evaluated this hypothesis.

As the subject is prepared for surgery 2 contact probes will be placed on the forehead to monitor the rSO2 and cerebral blood flow. This monitor can also measureblood flow velocity in blood vessels in the forehead.

This will only be done while the subject is on the cardiac bypass machine during the surgery and end shortly after entering the intensive care unit.Prior to surgery and then once a day on three of the first four postoperative days, patients will be assessed for the presence and severity of delirium with brief standard psychological exams. We will compare rSO2 and CBF changes between patients with and without delirium

ELIGIBILITY:
Inclusion Criteria:

* Patients in the study will be 50 or older undergoing elective cardiovascular surgery using cardiopulmonary bypass.
* Patients who can speak, read and understand the English language.
* Patients who understand the nature of the study and are willing to sign the consent form

Exclusion Criteria:

* Emergency surgery or patients intubated before surgery and, thus, cannot give informed consent.
* Patients diagnosed with neurocognitive disorders (e.g. Alzheimer's, Dementia)
* MMSE score greater than 21 Patients taking antipsychotic drugs A history of drug abuse
* Patients with an implant in the brain underneath the CerOx probes
* Women who are pregnant.
* History of significant, prohibitive skin allergies or reactions-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are under going cardiac bypass surgery with the use of cardiac perfusion
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To evaluate whether rSO2 and/or CBF during CPB is lower in patients who experience delirium within three days after cardiac surgery compared with patients without delirium | 3 days post op
  To evaluate whether rSO2 and/or CBF during CPB is lower in patients who experience delirium within three days after cardiac surgery compared with patients without delirium.

SECONDARY OUTCOMES:
recovery pattern of rSO2 | 3 post op days
  To evaluate the recovery pattern of rSO2 and CBF for up to 6 hrs after CPB for ICU patients who experience delirium within three days after cardiac surgery compared with patients without delirium.

OTHER OUTCOMES:
Can CBF autoregulation can be monitored using ultrasound compared with TCD | 3 days post op
  To assess whether CBF autoregulation can be monitored using ultrasound tagged light methodology compared with TCD
To evaluate the incidence of delirium in patients with impaired autoregulation | 3 days post op
  To evaluate the incidence of delirium in patients with impaired autoregulation

CONTACTS AND LOCATIONS:
Overall Officials: Kaushik Mandal, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States